CLINICAL TRIAL: NCT00014053
Title: A Study of Immune Function in Healthy Adults Aged 18-30 and 45 and Older
Brief Title: A Study of Immune System Activity in Healthy Adults
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG A5113; AACTG A5113
Record Dates: First submitted 2001-04-10; First posted 2001-08-31 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2003-06

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Reference Values; HIV Seropositivity; Immune System; CD4-Positive T-Lymphocytes; HIV Seronegativity; Antigens, CD
MeSH Terms: conditions — HIV Infections; HIV Seropositivity

SUMMARY:
The purpose of this study is to compare immune system activity in young people and older people who do not have HIV. This information will be compared to that of HIV patients in another study.

Aging affects immune system activity. This study will look at some of the factors involved. HIV also affects immune system activity. The results from this study, using healthy volunteers, will be compared to those in another study of HIV-infected patients. This may provide information on immune system activity in aging and HIV.

DETAILED DESCRIPTION:
Aging is associated with declines in both cellular and humoral immunity. A consistent observation of the aging immune system is a change in T cells. Another possible mechanism of diminished cellular immunity associated with age includes accelerated lymphocyte apoptosis. Enhanced lymphocyte apoptosis may play an important role in the pathogenesis of HIV disease. This study will use healthy volunteers to confirm and expand upon such observations. Samples from these volunteers will serve as controls to those from the HIV-infected participants of A5015 (a comparison study of 2 age-differentiated cohorts to determine potential mechanisms that might contribute to accelerated HIV-disease progression that is associated with aging).

This is a non-treatment study; however, volunteers receive hepatitis A and tetanus vaccinations. Numbers of phenotypically naive CD4+ cells (CD45RA+/CD62L+) are compared between healthy, HIV-seronegative volunteers and HIV-seropositive patients of A5015. An array of assays to assess baseline differences in immune function between these study populations are performed. Expression of markers of activation are compared by measuring the coexpression of HLA-DR+/CD38+ and CD28+ on CD4+ and CD8+ lymphocytes between these populations. To investigate possible age-associated differences in apoptosis, Fas (CD95+) expression is measured on CD4+ and CD8+ T cells by flow cytometry, and spontaneous apoptosis is assessed using the propidium iodide method. DTH hypersensitivity to skin test antigens, lymphocyte proliferation to mitogens, soluble antigens, recall antigens, and neoantigens are compared between the 2 populations. Antibody responses to vaccination with tetanus and hepatitis A are assessed. Finally, thymic size as measured by CT scan and the frequency of T cells that contain TRECs is compared between these 2 populations.

ELIGIBILITY:
Inclusion Criteria

Volunteers may be eligible for this study if they:

* Are willing to undergo HIV testing.
* Have a negative urine or serum pregnancy test within 30 days prior to study entry (for women volunteers).
* Are between the ages of 18 and 30 or are 45 or older.

Exclusion Criteria

Volunteers will not be eligible for this study if they:

* Have HIV infection.
* Have a serious infection or other serious medical illness that requires treatment and/or hospitalization within 90 days before study entry.
* Have had cancer.
* Have received any of the following within 6 months of study entry: systemic corticosteroids; chemotherapy or radiation; erythropoietin, granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), or growth hormone; drugs that affect the immune system including thalidomide, interleukins, interferons, or other cytokines; anabolic steroids at high levels; or any experimental agent, unless allowed otherwise by the researchers.
* Are immune to hepatitis A.
* Have received tetanus toxoid within 5 years prior to study entry or have a history of severe reaction to tetanus vaccine at any time in the past.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kalayjian, Study Chair
Locations (9):
- United States (9):
  - Univ of California San Francisco, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Washington Univ School of Medicine, St Louis, Missouri
  - Case Western Reserve Univ, Cleveland, Ohio
  - Univ of Texas Galveston, Galveston, Texas
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Derived] Tenorio AR, Spritzler J, Martinson J, Gichinga CN, Pollard RB, Lederman MM, Kalayjian RC, Landay AL. The effect of aging on T-regulatory cell frequency in HIV infection. Clin Immunol. 2009 Mar;130(3):298-303. doi: 10.1016/j.clim.2008.10.001. Epub 2008 Nov 12. PMID 19008157